CLINICAL TRIAL: NCT00001392
Title: Pathogenesis of Glomerulosclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940127; 94-DK-0127
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-17

CONDITIONS: Glomerular Disease
Keywords: Rituximab; Renal Biopsy; Viral Infection; Biomarkers; Natural History
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Subjects with known or suspected forms of sclerosing glomerular or chronic, fibrosing tubulointerstitial kidney diseases

SUMMARY:
The present protocol seeks to advance our understanding of sclerosing glomerular and tubulointerstitial kidney diseases, including but not limited to variants of focal segmental glomerulosclerosis (FSGS) and chronic kidney disease of unknown etiology (CKDu). This protocol will encompass studies of the natural history, pathogenesis and treatment of these chronic kidney disorders. It will also allow us to: (1) provide second opinions to referring physicians about management of subjects with these relatively rare kidney diseases; (2) collect research samples (e.g., blood), urine, and kidney tissue obtained from clinically-indicated or from research renal biopsies); (3) and treat these subjects with standard or other approved therapies; or (4) invite selected subjects patients to participate in limited pilot studies of novel combinations of standard therapeutic agents, such as rituximab and cyclosporine. (5) Agricultural worker chronic kidney disease of undetermined etiology (CKDu) is a growing problem in tropical countries in the Americas and Asia, including Sri Lanka where collaborators are located. We will receive kidney tissue from 25 CKDu cases for pathologic examination and transcriptional profiling and blood, plasma, serum, urine for metabolomic and genetic analysis from 50 cases and controls. Subjects were consented and samples were collected under a protocol approved by the University of Colombo IRB. These studies may provide the opportunity to generate new hypotheses regarding pathogenesis and treatment that would be candidates for testing in other research protocols.

Subjects with known or suspected forms of sclerosing glomerular or chronic, fibrosing tubulointerstitial kidney diseases will undergo routine medical evaluation, laboratory testing, imaging procedures and kidney biopsies as medically indicated. Selected subjects will be invited to provide informed consent to undergo a kidney biopsy for research purposes. Blood, urine, and tissue samples will be evaluated both for standard diagnostic purposes and for research purposes using specialized molecular methods that may provide insights into specific disease pathogenesis. Subjects may elect to receive the results of their kidney disease evaluation, NIH treatment recommendations, and return to the care of their referring physicians. Other subjects may be treated with either conventional or approved agents, or (with separate consent) with a novel combination of conventional therapies (rituximab and cyclosporine) as part of pilot studies that would involve long-term follow-up care at the NIH....

DETAILED DESCRIPTION:
The present protocol seeks to advance our understanding of sclerosing glomerular and tubulointerstitial kidney diseases, including but not limited to variants of focal segmental glomerulosclerosis (FSGS) and chronic kidney disease of unknown etiology (CKDu). This protocol will encompass studies of the natural history, pathogenesis and treatment of these chronic kidney disorders. It will also allow us to: (1) provide second opinions to referring physicians about management of subjects with these relatively rare kidney diseases; (2) collect research samples (e.g., blood), urine, and kidney tissue obtained from clinically-indicated or from research renal biopsies); (3) and treat these subjects with standard or other approved therapies; or (4) invite selected subjects patients to participate in limited pilot studies of novel combinations of standard therapeutic agents, such as rituximab and cyclosporine. (5) Agricultural worker chronic kidney disease of undetermined etiology (CKDu) is a growing problem in tropical countries in the Americas and Asia, including Sri Lanka where collaborators are located. We will receive kidney tissue from 25 CKDu cases for pathologic examination and transcriptional profiling and blood, plasma, serum, urine for metabolomic and genetic analysis from 50 cases and controls. Subjects were consented and samples were collected under a protocol approved by the University of Colombo IRB. These studies may provide the opportunity to generate new hypotheses regarding pathogenesis and treatment that would be candidates for testing in other research protocols.

Subjects with known or suspected forms of sclerosing glomerular or chronic, fibrosing tubulointerstitial kidney diseases will undergo routine medical evaluation, laboratory testing, imaging procedures and kidney biopsies as medically indicated. Selected subjects will be invited to provide informed consent to undergo a kidney biopsy for research purposes. Blood, urine, and tissue samples will be evaluated both for standard diagnostic purposes and for research purposes using specialized molecular methods that may provide insights into specific disease pathogenesis. Subjects may elect to receive the results of their kidney disease evaluation, NIH treatment recommendations, and return to the care of their referring physicians. Other subjects may be treated with either conventional or approved agents, or (with separate consent) with a novel combination of conventional therapies (rituximab and cyclosporine) as part of pilot studies that would involve long-term follow-up care at the NIH.

ELIGIBILITY:
* EVALUATION AND TREATMENT OF GLOMERULOSCLEROSIS
* INCLUSION CRITERIA:

  ---An unlimited number of subjects with known or suspected glomerular or tubulointerstitial disease will be eligible for study. No sex, race or ethnic selection will be applied. It is anticipated the African-Americans will predominate, given the increased risk of FSGS (focal segmental glomerulosclerosis) in this population.
* EXCLUSION CRITERIA:

  ---None

  -WHOLE EXOME/GENOME SEQUENCING
* ELIGIBLITY FOR WHOLE EXOME/GENOME SEQUENCING:

  * Subjects with kidney disease

    * Unexplained kidney disease, family history of kidney disease, or other kidney disease suggestive of a genetic origin, excluding FSGS
    * Age greater than or equal to 2 years
  * Subjects without kidney disease

    * Family member with unexplained kidney disease, family history of kidney disease, or other kidney disease suggestive of a genetic origin, excluding FSGS
    * Age greater than or equal to 18 years
    * Able to provide informed consent

      * RITUXIMAB AND CYCLOSPORINE. (CLOSED FOR SUBJECT RECRUITMENT.)
* INCLUSION CRITERIA FOR ADULT PATIENTS PARTICIPATING IN PILOT STUDY OF COMBINATION RITUXIMAB AND CYCLOSPORINE:

  * First void urine protein to creatinine ratio > 2g/g despite optimal use of an ACE inhibitor or ARB (or possibly both), last dose increase at least 4 weeks before qualifying proteinuria determination
  * Women must use reliable birth control method to avoid pregnancy while participating in the study.
  * Subjects who have failed to respond with a complete remission or partial remission after at least 8 weeks of prednisone at a dose of at least 60 mg or are steroid dependent or relapse off steroids.
  * Subjects who have compelling contraindications to the use of glucocorticoids, such as morbid obesity, defined as BMI >35 or diabetes mellitus
  * Subjects with idiopathic FSGS or collapsing glomerulopathy
  * Subjects with eGFR greater than or equal to 50 mL/min/1.73 m^2 at screening or at some time in preceding 6 months.
* INCLUSION CRITERIA FOR MINORS (BETWEEN AGES 4 AND 18 YEARS):

  * Estimated average protein to creatinine ratio >2.0 g/g despite use of an ACE inhibitor or ARB. At least one-first void urine will be obtained and must have a urine protein/creatinine ratio >2.0 g/g to exclude the diagnosis of orthostatic proteinuria
  * Girls who are going through puberty and/or have menstrual periods must use reliable birth control method to avoid pregnancy while participating in the study
  * Failed to respond with a complete remission or partial remission after at least 8 weeks of prednisone at a dose of at least 1 mg/kg or are steroid dependent or relapse off steroids.
  * Compelling contraindications to the use of glucocorticoids, such as morbid obesity, defined as 99th percentile for age and sex, or diabetes mellitus
  * Subjects with idiopathic FSGS or collapsing glomerulopathy
  * Subjects with eGFR greater than or equal to 50 mL/min/1.73 m^2 at screening or at some time in preceding 6 months.
* EXCLUSION CRITERIA:

  * Age < 4 years.
  * Prior intolerance of rituximab or other monoclonal antibody therapy, including severe infusion reaction or hypersensitivity to murine proteins.
  * History of cardiac arrhythmias, unless cardiology consult approves the use of rituximab.
  * Treatment with rituximab within the last two years.
  * Prior intolerance of cyclosporine.
  * Subjects with post-adaptive FSGS (including obesity-associated FSGS, reflux nephropathy, reduced nephron mass). There is not a strong rationale for the use of immunologic therapy in this population.
  * Subjects with genetic FSGS due to a high penetrance mutation, e.g. NPHS2 mutation. There is not a strong rationale for the use of immunologic therapy in this population.
  * Medication-associated FSGS.
  * Recurrent FSGS following renal transplant
  * Chronic viral infection, such as HIV-1, hepatitis B, and hepatitis C. The safety of aggressive immunologic therapy in these diseases is in question.
  * Chronic bacterial infection. At baseline, if the patient gives a history of BCG vaccination or prior positive PPD, we will consult with an infectious disease clinician before enrolling the patient.
  * Active malignancy
  * Poorly controlled hypertension is defined as home BP measurements >140/90 or controlled blood pressure requiring 4 or more medications. The rationale is that blood pressure elevation is common on cyclosporine therapy.
  * Women and girls who are pregnant or trying to become pregnant or are unwilling to practice birth control. Rituximab is in pregnancy class C: no systematic evidence of safety. In humans, cyclosporine crosses the placenta. Cyclosporine lacks genotoxic effects in human and animal studies. However, growth restriction and prematurity occur in up to 40% of neonates born to mothers with organ transplants who are treated with cyclosporine, but no congenital abnormalities have been documented.
  * Women and girls who are breastfeeding (possible immune suppression in infants as well as the unknown effects on growth or association with carcinogenesis.)
  * Predicted requirement for live vaccines over the 24 months following enrollment.

    * ANALYSIS OF LIPID-CONTAINING PARTICLES CHARACTERISTICS UNDER NUCLEAR MAGNETIC RESONANCE SPECTROSCOPY (NMR-S) AMONG NEPHROTIC SUBJECTS
* INCLUSION CRITERIA:

  * We will enroll adult subjects (greater than or equal to 18 years of age), male or female, and of all racial backgrounds/ethnicities. In this cohort, we will include subjects with kidney disease or without kidney disease (healthy volunteers). We will start with subjects with preserved glomerular filtration rate (eGFR-Cr greater than or equal to 60 ml/min/1.73m2) but may expand to include individuals with lower GFR in a later study. We will estimate glomerular filtration rate (eGFR) using the 2009 CKD-EPI creatinine equation.
  * In respect to proteinuria, we will accept both urine protein-to-creatinine ratio (uPCR) or urine protein excretion rate (PER) per 24 hours as a selection criteria. We will divide enrolled subjects in 3 groups as shown below:
  * Group 1. Subjects with nephrotic range proteinuria (uPCR greater than or equal to 2 g/g or PER greater than or equal to 3 gr/24hs.) and eGFR-Cr greater than or equal to 60 ml/min/1.73m2, regardless of their albumin levels.
  * Group 2. Subjects with sub-nephrotic range proteinuria (uPCR greater than or equal to 0.2 g/g but < 2 g/g or PER greater than or equal to 300 mg/24hs. but < 3 gr/24hs.) and eGFR-Cr greater than or equal to 60 ml/min/1.73m2, regardless of their albumin levels.
  * Group 3. Volunteers with normal eGFR and normal protein excretion and normal fasting clinical lipid testing.
  * For those subjects undergoing lipid lowering therapies for primary prevention, including statins, fibrates, niacin, ezetimibe, bile acid resins, fish oil or red yeast rice, we will stop those treatments at least 4 weeks but no more than 6 weeks prior their admission. Lipid lowering therapy will not be stopped for more than 8 weeks. We will not enroll subjects who are receiving statins or other lipid lowering therapies for secondary prevention. Also, we will not enroll subjects with history of triglycerides levels >1000 mg/dl.
  * The blood and urine sample collection and brief interruption of statin treatment performed in this pilot study to involve no more than minimal risk to individual subjects, with no prospect of direct benefit to subjects, but likely to yield generalizable knowledge to further society's understanding of the lipoprotein profiles of nephrotic and non-nephrotic subjects.
* EXCLUSION CRITERIA:

  * We will exclude subjects with any of the following:

    * Diabetes mellitus
    * Body mass index (BMI) greater than or equal to 40,
    * Pregnant or breastfeeding women
    * Untreated or uncontrolled thyroid disorder
    * Active oncologic condition
    * Acute infections
    * Chronic infections including HIV
    * Subjects receiving lipid lowering medications for secondary prevention (e.g. coronary artery disease, stroke, heart failure)
    * Subjects receiving estrogen therapy or contraceptive therapy
    * Subjects receiving cyclosporine, azathioprine or sirolimus
    * Subjects who are unable to eat the required meals due to allergy, intolerance, or dietary preferences
    * Subjects with history of pancreatitis
    * Subjects with reported history of triglycerides >1000 mg/dl
    * Subjects unable or unwilling to give their consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with known or suspected glomerular or tubulointerstitial disease will be eligible for study. No sex, race or ethnic selection will be applied. It is anticipated the African-Americans will predominate, given the increased risk of FSGS in this population. For evaluation, treatment, and pathogenetic studies, we will enroll children >=2 years of age and adults, including pregnant women and impaired subjects, if they have known or suspected forms of the kidney diseases described above. For pathogenetic studies not involving interventional procedures such as renal biopsies, we will also include healthy volunteers, including children >=12 years of age and adults. We will also recruit subjects including children >=12 years of age and adults with autoimmune and inflammatory diseases, both with and without kidney disease, to serve as controls for subjects with the sclerosing glomerular kidney diseases that are the primary focus of this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 537 (Actual)
Dates: Start 1996-04-16 (Actual)

PRIMARY OUTCOMES:
new hypotheses | one year
  To generate new hypotheses regarding pathogenesis and treatment that would be candidates for testing in other research protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Anirban Ganguli, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD is not consistent with the consents for this study. Data has been published in three peer-reviewed journal articles, listed here: @@@@@@Orloff MS, Iyengar SK, Winkler CA, Goddard KA, Dart RA, Ahuja TS, et al. Variants in the Wilms' tumor gene are associated with focal segmental glomerulosclerosis in the African American population. Physiol Genomics. 2005;21(2):212-21.@@@@@@Kopp JB, Smith MW, Nelson GW, Johnson RC, Freedman BI, Bowden DW, et al. MYH9 is a major-effect risk gene for focal segmental glomerulosclerosis. Nat Genet. 2008;40(10):1175-84.@@@@@@Genovese G, Friedman DJ, Ross MD, Lecordier L, Uzureau P, Freedman BI, et al. Association of trypanolytic ApoL1 variants with kidney disease in African Americans. Science. 2010;329(5993):841-5.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1994-DK-0127.html